CLINICAL TRIAL: NCT02142283
Title: Diffusion Weighted Imaging (DWI) or Computerized Tomography Perfusion (CTP) Assessment With Clinical Mismatch in the Triage of Wake Up and Late Presenting Strokes Undergoing Neurointervention (DAWN)
Brief Title: Clinical Mismatch in the Triage of Wake Up and Late Presenting Strokes Undergoing Neurointervention With Trevo
Acronym: DAWN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T4024
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Stroke
Keywords: Mechanical thrombectomy; Acute ischemic stroke; Wake up stroke; Late presenting stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trevo Thrombectomy Procedure (Experimental): Trevo Thrombectomy Procedure and Medical Management
  Interventions: Device: Trevo Thrombectomy Procedure; Other: Medical Management
- Medical Management (Active Comparator): Medical Management
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: Trevo Thrombectomy Procedure — stent retriever; intended to restore blood flow in the neurovasculature by removing thrombus (clot)
  Other Names: Trevo ProVue Retriever; Trevo XP ProVue Retriever
  Arms: Trevo Thrombectomy Procedure
Other: Medical Management — Standard of Care not including mechanical thrombectomy, no intra arterial treatment, may include aspirin, therapy etc
  Other Names: Standard of Care

SUMMARY:
The purpose of the study is to evaluate the hypothesis that Trevo thrombectomy plus medical management leads to superior clinical outcomes at 90 days as compared to medical management alone in appropriately selected subjects experiencing an acute ischemic stroke when treatment is initiated within 6-24 hours after last seen well.

DETAILED DESCRIPTION:
The study is a prospective, randomized, multi-center, Phase II/III (feasibility/pivotal), adaptive, controlled trial, designed to demonstrate that mechanical thrombectomy using the Trevo Retriever with medical management is superior to medical management alone in improving clinical outcomes at 90 days in appropriately selected wake up and late presenting acute ischemic stroke subjects.

The intent of this study is to support the use of the Trevo Retriever beyond the currently labeled 8 hour indicated time limit in wake up, unclear onset, and late presenting ischemic stroke subjects, who currently have no other option besides medical management of their symptoms.

Patients with wake-up strokes, strokes with unclear onset time, and witnessed late presenting strokes may potentially benefit from intra-arterial reperfusion therapy. However, an important indicator of whether subjects will benefit or not during this later time window is the confirmation of a large vessel occlusion (LVO), and assessment of the core infarct volume relative to the volume of salvageable penumbra. Therefore, standardized imaging selection of subjects is required for inclusion into the study.

This trial has been designed with subject safety in mind, as a seamless Phase II (feasibility) / Phase III (pivotal) adaptive design, in order to address the concerns around potential unknown harms to enrolled subjects. This study will help to answer the question of whether carefully selecting subjects by using Clinical Imaging Mismatch will allow acute ischemic stroke patients who present at or beyond 6 hours from Time Last Seen Well (TLSW) to be considered for intra-arterial intervention. If Trevo thrombectomy plus medical management leads to better clinical outcomes over medical management alone, more patients in the future could receive endovascular treatment (either in addition to or in lieu of IV tPA).

ELIGIBILITY:
General Inclusion Criteria:

1. Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke, and subject belongs to one of the following subgroups:

   1. Subject has failed IV t-PA therapy (defined as a confirmed persistent occlusion 60 min after administration)
   2. Subject is contraindicated for IV t-PA administration
2. Age ≥18
3. Baseline NIHSS ≥10 (assessed within one hour of measuring core infarct volume)
4. Subject can be randomized between with 6 to 24 hours after time last known well
5. No significant pre-stroke disability (pre-stroke mRS must be 0 or 1)
6. Anticipated life expectancy of at least 6 months
7. Subject willing/able to return for protocol required follow up visits
8. Subject or subject's Legally Authorized Representative (LAR) has signed the study Informed Consent form*

   * If approved by local ethics committee and country regulations, the investigator is allowed to enroll a patient utilizing emergency informed consent procedures if neither the patient nor the representative or person of trust is available to sign the informed consent form. However, as soon as possible, the patient is informed and his/her consent is requested for the possible continuation of this research. (Not applicable to U.S. Sites.)

Imaging Inclusion Criteria:

1. < 1/3 MCA territory involved, as evidenced by CT or MRI
2. Occlusion of the intracranial ICA and/or MCA-M1 as evidenced by MRA or CTA
3. Clinical Imaging Mismatch (CIM) defined as one of the following on MR-DWI or CTP-rCBF maps:

   1. 0-<21 cc core infarct and NIHSS ≥ 10 (and age ≥ 80 years old)
   2. 0-<31 cc core infarct and NIHSS ≥ 10 (and age < 80 years old)
   3. 31 cc to <51 cc core infarct and NIHSS ≥ 20 (and age < 80 years old)

General Exclusion Criteria:

1. History of severe head injury within past 90 days with residual neurological deficit, as determined by medical history
2. Rapid improvement in neurological status to an NIHSS <10 or evidence of vessel recanalization prior to randomization
3. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept)
4. Seizures at stroke onset if it makes the diagnosis of stroke doubtful and precludes obtaining an accurate baseline NIHSS assessment
5. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol)
6. Baseline hemoglobin counts of <7 mmol/L
7. Baseline platelet count < 50,000/uL
8. Abnormal baseline electrolyte parameters as defined by sodium concentration <130 mmol/L, potassium concentration <3 mEq/L or >6 mEq/L
9. Renal failure as defined by a serum creatinine >3.0 mg/dL (264 µmol/L) NOTE: subjects on renal dialysis may be treated regardless of serum creatinine levels
10. Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with INR > 3.0 or PTT > 3 times normal. Patients on factor Xa inhibitor for 24-48 hours ago must have a normal PTT.
11. Any active or recent hemorrhage within the past 30 days
12. History of severe allergy (more than rash) to contrast medium
13. Severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using medication the subject can be enrolled
14. Female who is pregnant or lactating at time of admission
15. Current participation in another investigational drug or device study
16. Presumed septic embolus, or suspicion of bacterial endocarditis
17. Treatment with any cleared thrombectomy devices or other intra-arterial (neurovascular) therapies prior to randomization

Imaging Exclusion Criteria:

1. Evidence of intracranial hemorrhage on CT/MRI
2. CTA or MRA evidence of flow limiting carotid dissection, high-grade stenosis, or complete cervical carotid occlusion requiring stenting at the time of the index procedure (i.e., mechanical thrombectomy).
3. Excessive tortuosity of cervical vessels on CTA/MRA that would likely preclude device delivery/deployment
4. Suspected cerebral vasculitis based on medical history and CTA/MRA
5. Suspected aortic dissection based on medical history and CTA/MRA
6. Intracranial stent implanted in the same vascular territory that would preclude the safe deployment/removal of the Trevo device
7. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior circulation/vertebrobasilar system) as confirmed on CTA/MRA, or clinical evidence of bilateral strokes or strokes in multiple territories
8. Significant mass effect with midline shift as confirmed on CT/MRI
9. Evidence of intracranial tumor (except small meningioma) as confirmed on CT/MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-07; Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tudor G Jovin, MD, Principal Investigator — University of Pittsburg Medical Center Stroke Institute; Raul Nogueira, MD, Principal Investigator — Marcus Stroke & Neuroscience Center, Grady Memorial Hospital
Locations (32):
- United States (24):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Christiana Care, Newark, Delaware
  - Memorial Regional, Hollywood, Florida
  - Baptist Jacksonville, Jacksonville, Florida
  - Jackson Memorial/University of Miami, Miami, Florida
  - Florida Hospital; Neuroscience Research Center, Orlando, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - RUSH University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - St. Joseph Mercy - Oakland, Pontiac, Michigan
  - JFK Neuroscience Institute at JFK Medical Center, Edison, New Jersey
  - Capital Health System, Trenton, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital/ Ohio Health Research Institute, Columbus, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Stroke Institute, Pittsburgh, Pennsylvania
  - Erlanger Health System, Chattanooga, Tennessee
  - Valley Baptist Medical Center-Harlingen, Harlingen, Texas
  - North Texas Stroke Center HCA (dba TSI), Plano, Texas
- Royal Melbourne, Parkville, Australia
- Toronto Western Hospital - University Health Network, Toronto, Ontario, Canada
- France (2):
  - Hôpital Gui de Chauliac, Montpellier
  - Hopital Purpan - Toulouse, Toulouse
- Spain (4):
  - Vall d'Hebron Barcelona, Barcelona
  - Hospital Clinic - Barcelona, Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona

REFERENCES:
- [Derived] Roaldsen MB, Lindekleiv H, Mathiesen EB. Intravenous thrombolytic treatment and endovascular thrombectomy for ischaemic wake-up stroke. Cochrane Database Syst Rev. 2021 Dec 1;12(12):CD010995. doi: 10.1002/14651858.CD010995.pub3. PMID 34850380
- [Derived] Liebeskind DS, Saber H, Xiang B, Jadhav AP, Jovin TG, Haussen DC, Budzik RF, Bonafe A, Bhuva P, Yavagal DR, Hanel RA, Ribo M, Cognard C, Sila C, Hassan AE, Smith WS, Saver JL, Nogueira RG; DAWN Investigators. Collateral Circulation in Thrombectomy for Stroke After 6 to 24 Hours in the DAWN Trial. Stroke. 2022 Mar;53(3):742-748. doi: 10.1161/STROKEAHA.121.034471. Epub 2021 Nov 3. PMID 34727737
- [Derived] Liebeskind DS, Saber H, Bhuva P, Xiang B, Yoo AJ, Jadhav AP, Haussen DC, Budzik RF, Bonafe A, Yavagal DR, Hanel RA, Ribo M, Cognard C, Sila C, Hassan AE, Smith WS, Saver JL, Nogueira RG, Jovin TG. Serial ASPECTS in the DAWN Trial: Infarct Evolution and Clinical Impact. Stroke. 2021 Oct;52(10):3318-3324. doi: 10.1161/STROKEAHA.120.033477. Epub 2021 Jul 20. PMID 34281376
- [Derived] Tekle WG, Hassan AE, Jadhav AP, Haussen DC, Budzik RF, Bonafe A, Bhuva P, Yavagal DR, Hanel RA, Ribo M, Cognard C, Sila CA, Smith WS, Saver JL, Liebeskind DS, Shields R, Nogueira RG, Jovin TG; DAWN Trial Investigators. Impact of Periprocedural and Technical Factors and Patient Characteristics on Revascularization and Outcome in the DAWN Trial. Stroke. 2020 Jan;51(1):247-253. doi: 10.1161/STROKEAHA.119.026437. Epub 2019 Nov 20. PMID 31744425
- [Derived] Aghaebrahim A, Jadhav AP, Hanel R, Sauvageau E, Granja MF, Zhang Y, Haussen DC, Budzik RF, Bonafe A, Bhuva P, Ribo M, Cognard C, Sila C, Yavagal D, Hassan AE, Smith WS, Saver J, Liebeskind DS, Nogueira RG, Jovin TG; DAWN Investigators. Outcome in Direct Versus Transfer Patients in the DAWN Controlled Trial. Stroke. 2019 Aug;50(8):2163-2167. doi: 10.1161/STROKEAHA.119.025710. Epub 2019 Jul 15. PMID 31303153
- [Derived] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: See protocol
Pre-assignment Details: See protocol
Period: Overall Study
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Started | 107 | 99
Completed | 86 | 78
Not Completed | 21 | 21
Not completed — Death | 20 | 18
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Trevo Thrombectomy Procedure | Medical Management | Total
Number analyzed (Participants) | 107 | 99 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.4 (14.1) | 70.7 (13.2) | 70.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 48 | 113
  Male | 42 | 51 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 27
  Not Hispanic or Latino | 94 | 82 | 176
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 23 | 15 | 38
  White | 70 | 63 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Weighted Modified Rankin Scale (mRS) Score, Lead Co-Primary Efficacy Outcome
Description: mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes neurological disability.
  Functional Independence:
  0 - no symptoms at all
  1. - no significant disability despite symptoms; able to carry out all usual duties and activities
  2. - slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - moderate disability; requiring some help, but able to walk without assistance
  4. - moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - dead
Time Frame: 90 days
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
score on a scale | 5.5 (3.8) | 3.4 (3.2)

2. Primary Outcome: Functional Independence (mRS 0-2), Nested Co-Primary Efficacy Outcome
Description: Number of participants with functional independence
  mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes neurological disability.
  Functional Independence:
  0 - no symptoms at all
  1. - no significant disability despite symptoms; able to carry out all usual duties and activities
  2. - slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
Time Frame: 90 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 52 | 13

3. Primary Outcome: Stroke-related Mortality, Primary Safety Outcome
Time Frame: 90 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 17 | 18

4. Secondary Outcome: Good Functional Outcome
Description: Proportion of participants with functional independence
  mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes neurological disability.
  Functional Independence:
  0 - no symptoms at all
  1. - no significant disability despite symptoms; able to carry out all usual duties and activities
  2. - slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
Time Frame: 90 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 52 | 13

5. Secondary Outcome: Early Response
Description: The proportion of subjects with "early response" at Day 5-7/Discharge (whichever is earlier), defined as a National Institutes of Health Stroke Scale (NIHSS) drop of ≥10 from baseline or NIHSS score 0 or 1.
  The NIHSS is an assessment which objectively quantifies the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Time Frame: 5-7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 51 | 19

6. Secondary Outcome: All Cause Mortality
Time Frame: 90 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 20 | 18

7. Secondary Outcome: Revascularization Rates
Description: Revascularization rates at 24 hours from randomization are based on the assessment of vessel patency utilizing CTA/MRA and processed by the CT-MR core laboratory. Revascularization at 24 hours was defined as the presence of partial or complete recanalization.
  CTA/MRA images utilized ionizing radiation exposure.
Time Frame: 24 hours
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 82 | 38

8. Secondary Outcome: Neurological Deterioration From Baseline NIHSS Score
Description: Neurological deterioration from baseline NIHSS score through Day 5-7/discharge (whichever is earlier) post randomization. Neurological deterioration is defined as ≥ 4 point increase in the NIHSS score from the baseline score.
  The calculated difference in NIHSS scores was assessed at baseline and Day 5-7/discharge (two time points).
  The NIHSS is an assessment which objectively quantifies the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Time Frame: 5-7 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
Number analyzed (Participants) | 107 | 99
Participants | 15 | 26

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Trevo Thrombectomy Procedure | Medical Management
All-Cause Mortality (participants affected / at risk) | 20/107 | 18/99
Serious Adverse Events (participants affected / at risk) | 41/107 | 47/99
Other Adverse Events (participants affected / at risk) | 102/107 | 91/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trevo Thrombectomy Procedure (N=107) | Medical Management (N=99)
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pulmonary oedema (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 9
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Immune system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal pain (Injury, poisoning and procedural complications) | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0
Brain herniation (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 2 | 5
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Convulsion (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 3 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Muscular weakness (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 9
Status epilepticus (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 5 | 9
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Tracheal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Amputation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 2 | 1
Shock (Vascular disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Cranioplasty (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trevo Thrombectomy Procedure (N=107) | Medical Management (N=99)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 14 | 13
Bradycardia (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Pulmonary oedema (Cardiac disorders) | 3 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 4
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distention (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Clostridium difficile colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 10 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 7 | 13
Gastric hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hiccups (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 3
Chest pain (General disorders) | 1 | 0
Device occulsion (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Local swelling (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 6 | 8
Pyrexia (General disorders) | 8 | 5
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 2
Mucosal infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 3 | 3
Penumonia (Infections and infestations) | 6 | 8
Purulent discharge (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 2
Skin candida (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 22 | 22
Urosepsis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Nephropathy toxic (Injury, poisoning and procedural complications) | 1 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood lactate dehydrogenase abnormal (Injury, poisoning and procedural complications) | 1 | 0
Blood lactic acid increased (Injury, poisoning and procedural complications) | 0 | 1
Cardiac enzymes increased (Injury, poisoning and procedural complications) | 0 | 1
Computerised tomogram abnormal (Investigations) | 1 | 0
Electroencephalogram abnormal (Investigations) | 2 | 0
International normalized ratio increased (Investigations) | 0 | 1
Investigation abnormal (Investigations) | 0 | 1
Liver function analyses (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Troponin increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercreatinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypergylcaemia (Metabolism and nutrition disorders) | 7 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 2
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Monoarthritis (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Allodynia (Nervous system disorders) | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain herniation (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 5 | 7
Carotid artery stenosis (Nervous system disorders) | 3 | 1
Central pain syndrome (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 4 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischemia (Nervous system disorders) | 1 | 0
Cerebral microhemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 3
Confusional state (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 2
Cytotoxic edema (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2
Dysarthria (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 4
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 5 | 3
Haemorrhagic tranformation stroke (Nervous system disorders) | 25 | 16
Headache (Nervous system disorders) | 11 | 14
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 3
Muscular weakness (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Neurogenic bladder (Nervous system disorders) | 0 | 1
Neurogenic bowel (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 6 | 9
Neurological symptom (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Restless leg syndrome (Nervous system disorders) | 0 | 1
Restlessness (Nervous system disorders) | 1 | 0
Sleep apnoea syndrome (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 3 | 5
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 6 | 6
Anxiety (Psychiatric disorders) | 2 | 2
Anxiety disorder (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 4
Depressed mood (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 6 | 12
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 4
Mental status change (Psychiatric disorders) | 1 | 0
Somnolence (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 7
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 6 | 9
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 0 | 1
Penis disorder (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Aspiratoin (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Artial flutter (Cardiac disorders) | 2 | 1
Artial tachycardia (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Reaction to drug (Immune system disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter management (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Tumour excision (Surgical and medical procedures) | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 3
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 9 | 8
Hypotension (Vascular disorders) | 15 | 8
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral coldness (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 3
Vascular dissection (Vascular disorders) | 1 | 0
Vasospasm (Vascular disorders) | 3 | 0
Vessel puncture site haemorrhage (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall not make any publication without providing Sponsor 60 days notice. If Sponsor determines that the proposed publication contains confidential information, Sponsor may require the delay of publication for a period of time not to exceed 90 days and may require that any confidential information be removed from the publication. Sponsor may also require Physician to delay publication until any factual errors or inaccuracies in the publication are corrected.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT02142283/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02142283/SAP_001.pdf